CLINICAL TRIAL: NCT04148066
Title: Track and Treat in NSCLC (TATIN) - ctDNA Guided Treatment of Early Resistance to Targeted Treatment in Patients With EGFR Positive NSCLC
Brief Title: ctDNA Guided Treatment of Early Resistance to Targeted Treatment
Acronym: TATIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18TAT
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib and Crizotinib (Other): Osimertinib will be administered according to label: 80 mg once daily.
  Crizotinib will only be prescribed upon detection of MET amplification using ctDNA. Crizotinib will be administered according to label: 250 mg bi-daily.
  Interventions: Diagnostic Test: ctDNA blood sample

INTERVENTIONS:
Diagnostic Test: ctDNA blood sample — every six weeks during treatment and upon radiological progression blood will be drawn to analyse ctDNA with Avenio ctDNA (Expanded panel) to detect all known EGFR TKI resistance mechanisms.

SUMMARY:
The current strategy is to test for treatment resistance at the time of radiological progression and design subsequent treatment based on the mechanism of resistance. However, upon disease progression patients tend to deteriorate quickly and 30% - 40% of patients will not be in the clinical condition to receive next line treatment. Therefore, there is a potential for early resistance identification and directing treatment against it in order to improve patient outcome.

DETAILED DESCRIPTION:
Next Generation Sequence (NGS) technology rapidly evolves and it is now feasible to use circulating tumor DNA (ctDNA) as a BioSource for comprehensive analysis of the molecular make up of tumors. ctDNA based techniques are able to detect the emergence of drug resistance mechanisms with high sensitivity and prior to radiological progression (12-14). This technique might identify drug resistant clones before subclonal resistance (resistance of the new clone to targeted treatment) develops and allow to eliminate the new clone with short-term additional treatment, while continuing treatment of the main oncogenic driver (EGFR exon 19 del / exon 21 L858R) with the EGFR TKI. Continuous ctDNA based monitoring will reveal the success of the additional treatment and in case the follow-up ctDNA sample shows elimination of the EGFR TKI resistant clone, the add-on treatment will be discontinued. Continuous ctDNA based monitoring might identify a new resistant clone at a later point in time and temporary treatment of this clone can be initiated. The EGFR TKI will remain the backbone of therapy and will not be discontinued (see treatment strategy 1 in Figure 3).

This continuous track and treat strategy could potentially lead to a better outcome. In this study the investigators will track all known EGFR TKI resistance mechanisms over time and select one (MET amplification) for the track and treat strategy.

Treatment strategy 1: Track and treat strategy. ctDNA based resistance monitoring. As soon as a resistant clone is detected with ctDNA, treatment will be added to the EGFR TKI. ctDNA will be continuously screened for resistant clones. Upon disappearance of the resistant clone, add-on treatment will be discontinued, while the EGFR TKI will be continued at any time. Multiple resistance mechanisms can be treated serially.

Treatment strategy 2: routine care. Treatment with an EGFR TKI will be continued until radiological progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic NSCLC, characterized by a sensitizing exon 19 deletion or exon 21 L858R EGFR mutation.
2. WHO performance status 0-2.
3. Eligible for osimertinib treatment according to the label and according to the treating physician.
4. Patients must be ≥18 years of age.

Exclusion Criteria:

1. Patients with symptomatic central nervous system metastases who are neurologically unstable. Unstable brain metastases except for those who have completed definitive therapy and have had a stable neurological status for 2 weeks after completion of definitive therapy. Patients may be on corticosteroids to control brain metastases if they have been on a stable dose for 2 weeks prior to the start of study treatment and are clinically asymptomatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
percentage of patients in which a drug resistant clone can be detected with ctDNA | Trough study completion, an average of 2 years
  To identify the percentage of patients in which a drug resistant clone can be detected with ctDNA before the emergence of radiological progression.

SECONDARY OUTCOMES:
the success rate of crizotinib and osimertinib combination treatment to eliminate MET amplification | Trough study completion, an average of 2 years
  To determine the success rate of crizotinib and osimertinib combination treatment to eliminate MET amplification, defined by disappearance of the MET amplification clone in a subsequent ctDNA sample.

CONTACTS AND LOCATIONS:
Overall Officials: J de Langen, MD, PhD, Principal Investigator — The Netherlands Cancer Institute-Antoni van Leeuwenhoek
Locations (2):
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni van Leeuwenhoek, Amsterdam, North Holland
  - Erasmus MC, Universitair Medisch Centrum Rotterdam, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided